CLINICAL TRIAL: NCT05073419
Title: Arrhythmia Detection After Myocardial Infarction Trial
Brief Title: Arrhythmia Detection After MI
Acronym: AID MI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Samir Saba (Other)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor-Investigator, Samir Saba, Division Chief of Cardiology, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY21060027
Record Dates: First submitted 2021-09-28; First posted 2021-10-11 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Acute Myocardial Infarction
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Pilot randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Clinical information regarding ICM implantation will be withheld from outcome assessors
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Control (Active Comparator): Post-AMI patients in this arm will receive standard of care
  Interventions: Other: Standard of Care
- ICM (Experimental): Post-AMI patients in this arm will receive standard of care and an ICM
  Interventions: Device: ICM Implantation

INTERVENTIONS:
Other: Standard of Care — Routine monitoring of post AMI patient with clinic visits
  Other Names: Control
  Arms: Control
Device: ICM Implantation — Implantation of ICM through small incision (2 mm) under the skin
  Other Names: ICM
  Arms: ICM

SUMMARY:
Patients post acute myocardial infarction (AMI) have a high risk of mortality but the use of an implantable defibrillator in the early aftermath of an AMI has not been shown to improve patients' survival. The VEST trial recently demonstrated an improved overall survival in post AMI patients with the use of a wearable defibrillator. The same improvement was not demonstrated for the risk of sudden cardiac death. Monitoring patients after AMI using an implantable cardiac monitor (ICM) may document findings that can impact patient management and eventually improve their outcomes. We are therefore conducting the AID MI trial to examine the impact of ICM on patient management in the post AMI setting.

DETAILED DESCRIPTION:
Patients who have ventricular tachycardia or fibrillation at least 48 hours after an acute myocardial infarction (AMI) have a higher risk of sudden cardiac death. Current guidelines recommend that for primary prevention of sudden cardiac death, patients with left ventricular ejection fraction (LVEF) ≤ 35% should wait at least 40 days post-AMI or 90 days post revascularization prior to receiving an implantable cardioverter defibrillator (ICD). This period of time potentially leaves a vulnerable population without protection from sudden cardiac death (SCD).

The landmark MADIT I and MADIT II trials demonstrated that ICD therapy was associated with significantly improved survival in patients with ischemic cardiomyopathy at any interval of time. The DINAMIT study demonstrated that ICD placement less than 40 days after AMI had a reduction in arrhythmic mortality at the cost of an increase in non-arrhythmic mortality. Results from these and other studies suggest that the risk of SCD after AMI may be time-dependent and that patients at increased risk for SCD are also at increased risk for death from other causes. Thus, there is a need for additional studies to identify subsets of patients with arrhythmias that may benefit from other therapeutic interventions such as ablations, anti-arrhythmic medications, implantable cardiac devices, or other therapies.

The CARISMA study was the first study to document the incidence of cardiac arrhythmias in post-AMI patients with left ventricular dysfunction (LVEF≤40%) using an implantable loop recorder. Results showed high incidences of arrhythmias such as new-onset AF (27.6%) and high-degree AV block (9.8%). Subsequent studies showed that these arrhythmias were associated with increased risk of major cardiovascular events such as heart failure, ventricular tachyarrhythmias, stroke, reinfarction, or cardiac death.

It has been shown that utilizing remote monitoring as part of clinical care in patients with cardiac implantable electronic devices is associated with improved all-cause survival; the magnitude of survival increases with the degree of adherence to remote monitoring and the timeliness to enroll and activate in remote monitoring shortly after device implantation.

These studies suggest the need for further investigation and evaluation of acute and long-term cardiac monitoring in post-AMI patients, in an effort to identify patients at greatest risk, inform clinical decision making and potentially reduce the risk of all-cause mortality. In addition, the ability to remotely monitor patients may minimize the time to diagnosis and enable early intervention in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Adults, age 18 years or older
* AMI (STEMI and NSTEMI)
* Willing to give written informed consent
* Expected discharge from hospital within 7 days of AMI
* Willing to receive ICM insertion within 21 days of index AMI

Exclusion Criteria:

* Existing pacemaker, ICD, ICM, or any other implantable cardiac electronic device
* Pregnant
* Index AMI was more than 21 days
* Unwilling/cannot insert ICM within 21 days post AMI
* Planned ICD implant, planned CABG or any open-heart surgery (e.g. for severe valvular disease)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-08-09 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Changes to patient management | 90 days post AMI
  Incidence (frequency) of cardiac arrhythmias (bradyarrhythmia, tachyarrhythmia, pause, etc…) that lead to actionable treatment change
Time to diagnosis and/or treatment of cardiac arrhythmia | 90 days post AMI
  days post randomization

SECONDARY OUTCOMES:
Changes to patient management | 24 months
  Incidence (frequency) of cardiac arrhythmias (bradyarrhythmia, tachyarrhythmia, pause, etc…) that lead to actionable treatment change
Mortality | at 90 days
  all-cause mortality
Mortality | at 24 months
  All-cause mortality

OTHER OUTCOMES:
Depression and Anxiety Scale | at 90 days
  Hospital Anxiety and Depression Scale (HADS) Minimum 0 and maximum 21 0-7 = Normal 8-10 = Borderline abnormal (borderline case) 11-21 = Abnormal (case)
Depression and Anxiety Scale | at 24 months
  Hospital Anxiety and Depression Scale (HADS) Minimum 0 and maximum 21 0-7 = Normal 8-10 = Borderline abnormal (borderline case) 11-21 = Abnormal (case)
Physical and Mental Health | at 90 days
  PROMIS-29 scale Scale ranges from 29 to 145 with a higher number indicating better physical and mental health
Physical and Mental Health | at 24 months
  PROMIS-29 scale Scale ranges from 29 to 145 with a higher number indicating better physical and mental health

CONTACTS AND LOCATIONS:
Overall Officials: Samir F Saba, MD, Principal Investigator — University of Pittsburgh Medical Center
Locations (1):
- UPMC Presbyterian Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Publication of protocol, methods, results in aggregates
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 1 year after publication of the mainmanuscript
Access Criteria: Submit request to PI Only de-identified data will be shared